CLINICAL TRIAL: NCT01781338
Title: Adjuvant Dynamic Marker-Adjusted Personalized Therapy Trial Optimizing Risk Assessment and Therapy Response Prediction in Early Breast Cancer
Acronym: ADAPT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WSG-AM06 / ADAPT
Record Dates: First submitted 2013-01-25; First posted 2013-02-01 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction Therapy (Experimental): The kind of induction therapy is dependent on the respective sub-protocol.
  Interventions: Other: Induction therapy

INTERVENTIONS:
Other: Induction therapy — The intervention is dependent on the respective sub-protocol and can include either endocrine therapy, neoadjuvant chemotherapy or targeted therapy.

SUMMARY:
Trial for the optimization of risk assessment and therapy success prediction in patients with early breast cancer by the use of biomarkers in advance to therapy decision-making to personalize therapies.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age at diagnosis 18 years and above (consider patients at 70 years and above for ADAPT Elderly)
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Clinical T1 - T4 (except inflammatory breast cancer)
* All clinical N (cN)
* No clinical evidence for distant metastasis (M0)
* Known HR status and HER2 status (local pathology)
* Tumor block available for central pathology review
* Performance Status ECOG <= 1 or KI >= 80%
* Negative pregnancy test (urine or serum) within 7 days prior to start of induction treatment in premenopausal patients
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* The patient must be accessible for treatment and follow-up

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin or pTis of the cervix uteri
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
* Concurrent treatment with other experimental drugs. Participation in another interventional clinical trial with or without any investigational not marketed drug within 30 days prior to study entry
* Male breast cancer
* Concurrent pregnancy; patients of childbearing potential must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
* Breast feeding woman
* Sequential breast cancer
* Reasons indicating risk of poor compliance
* Patients not able to consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4936 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Identification of a responder sub-population with intermediate and high risk, which due to therapy has outcome comparable to HR+/RS≤11 | 8 years
  In order to identify patients that are at comparable low risk as hormone receptor positive, HER2 negative patients with low Recurrence Score, any sub-population across the sub-trials will be compared to this risk group.

SECONDARY OUTCOMES:
Overall survival | 8 years

OTHER OUTCOMES:
Any pre-specified outcome measure is defined within the sub-protocols. | 8 years
  Toxicity and cost efficacy are common endpoints of all sub-protocols. Additional "translational research" questions occurring during the trial will be defined in sub-protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Breast Center of the University of Munich (LMU) Universitätsfrauenklinik Großhadern, Munich, Germany; Ulrike Nitz, Prof. Dr., Study Chair — Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, Germany
Locations (2):
- Germany (2):
  - Breast Center of the University of Munich (LMU) Universitätsfrauenklinik Großhadern, Munich, Bavaria
  - Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, North Rhine-Westphalia

REFERENCES:
- [Background] Hofmann D, Nitz U, Gluz O, Kates RE, Schinkoethe T, Staib P, Harbeck N. WSG ADAPT - adjuvant dynamic marker-adjusted personalized therapy trial optimizing risk assessment and therapy response prediction in early breast cancer: study protocol for a prospective, multi-center, controlled, non-blinded, randomized, investigator initiated phase II/III trial. Trials. 2013 Aug 19;14:261. doi: 10.1186/1745-6215-14-261. PMID 23958221